CLINICAL TRIAL: NCT00038545
Title: A Phase II Study of Paclitaxel and Topotecan With Filgrastim-SD/01 Support For Patients With Relapsed and Refractory Aggressive Non-Hodgkin's Lymphoma
Brief Title: A Phase II Study of Paclitaxel and Topotecan With Filgrastim-SD/01 Support For Relapsed and Refractory Aggressive Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM01-008
Record Dates: First submitted 2002-05-31; First posted 2002-06-03 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: LYMPHOMA; NON-HODGKINS; AGGRESSIVE; RELAPSED AND REFRACTORY
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma; Aggression | interventions — pegfilgrastim; Paclitaxel; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Filgrastim SD/01
Drug: Paclitaxel
Drug: Topotecan

SUMMARY:
For patients with relapsed and refractory aggressive non-Hodgkin's lymphoma

ELIGIBILITY:
INCLUSION:

* Bidimensionally measurable current/refractory aggressive NHL (Diffuse lg cell, diffuse mixed cell, follicular lg non-cleaved, immunoblastic, Ki-1+ALCL, peripheral T-cell lymphoma, mantle cell lymphoma & transformed lymphoma.)
* No more than 3 prior treatment regimens. No anti-lymphoma therapy within the past 3 weeks.
* Not be eligible for treatment of a higher priority.
* Performance status <2 Zubrod, > 60 Karnofsky.
* Good marrow reserve: ANC>1.5 x 10(9)/L, platelets > 100 x 10(9)/L.
* Bilirubin <1.5mg/dL, SGOT, SGPT < 2 x normal values.
* Serum creatinine < 1.8 mg/dL.
* Age > 18 yrs.
* Signed informed consent.
* Life expectancy of > 12 weeks.
* No prior Taxane (paclitaxel or docetaxel), topotecan, or CPT-11.
* No prior stem cell or bone marrow transplantation.
* No prior second malignancies except for basal cell carcinoma of the skin.

EXCLUSION:

* Active or prior history of CNS lymphoma.
* Serious intercurrent medical illnesses requiring hospitalization.
* History of primary/secondary immunodeficiency (other than related to the malignant lymphoma because treatment is dependent on a functional immune system) or patients taking immunosuppressive drugs (systemic corticosteroids).
* Prior exposure to Filgrastim-SD/01.
* Women who are pregnant or lactating.
* Participation in another clinical trial.
* Positive HIV antibody.
* History of prior sensitivity to E. coli derived products (such as filgrastim/neupogen).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2001-05-18; Primary Completion 2004-04-27 (Actual); Study Completion 2004-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anas Younes, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States